CLINICAL TRIAL: NCT02838758
Title: A 3-arm Randomized Controlled Study Comparing Ultrasound-guided Cryoablation, Ultrasound-guided Perineural Lidocaine and Ultrasound-guided Perineural Saline to Treat Intermetatarsal Neuroma
Brief Title: Compare Ultrasound Assisted Cold Therapy and Lidocaine Injection to Treat Morton's Neuroma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, David Spinner, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 16-1139
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Intermetatarsal Neuroma
Keywords: Morton's neuroma; Intermetatarsal neuroma; forefoot pain; ultrasound guided cryoablation; ultrasound guided perineural lidocaine injection
MeSH Terms: conditions — Morton Neuroma | interventions — Cryosurgery; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cryoablation (Experimental): Ultrasound guided perineural cryoablation. The mechanism of therapeutic cryoablation involves using short and repeated cycles of freezing and thawing to cause axonal degeneration and disrupt neuronal activity without damage to epineurium and perineurium.
  Interventions: Device: Cryoablation
- Lidocaine (Active Comparator): Ultrasound guided perineural lidocaine injection. Under ultrasound guidance, roughly 3cc of 2% lidocaine will be injected near the neuroma.
  Interventions: Drug: Lidocaine
- Saline (Placebo Comparator): Ultrasound guided perineural normal saline injection. Under ultrasound guidance, roughly 3cc of normal saline will be injected near the neuroma.
  Interventions: Drug: Saline

INTERVENTIONS:
Device: Cryoablation — A minimally invasive cryoablation device. It delivers focused nitrous oxide to the target tissue via a 22-gauge needle to create an approximately 9.4mm by 5.4mm spherical freezing zone of temperature between -20 to -100° C.
  Other Names: Iovera
  Arms: Cryoablation
Drug: Lidocaine — Roughly 3cc of lidocaine will be injected near the intermetatarsal neuroma under ultrasound visualization.
  Other Names: xylocaine
  Arms: Lidocaine
Drug: Saline — Roughly 3cc of saline will be injected near the intermetatarsal neuroma under ultrasound visualization.
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a device that delivers freezing temperature compared to injecting lidocaine (an anesthetic medication) in providing pain relief to patients with disorganized nerve bundle between the toes, also known as Morton's neuroma. The same ultrasound technology that the obstetricians use to visualize a fetus inside a pregnant woman will be used to help the study physician to locate the Morton's neuroma while precisely delivering the freezing temperature and lidocaine near the nerve.

DETAILED DESCRIPTION:
This study will be a 3-arm randomized single-blinded placebo controlled study in which human subjects with intermetatarsal neuralgia will receive subcutaneous normal saline or subcutaneous lidocaine or ultrasound guided cryoablation. The first follow up will take place 4 weeks post procedure to monitor the magnitude and duration of pain relief. Subjects will then be crossed over. Those who had received saline or lidocaine will receive ultrasound guided cryoablation. Individuals, who had previously been given ultrasound guided cryoablation without any improvement, may opt for another denervation procedure at 4 weeks. All of the participants will be followed up at 3 months post procedure to determine the magnitude and duration of pain relief.

Study procedures will be conducted by the principle investigator who is a Board Certified pain management attending physician and an expert in performing ultrasonography guided interventions The cryoablation device is routinely used to treat various painful pathologies at Mount Sinai and Beth Israel pain management offices. The device manual and instructions will be available at both locations. All research staff has prior experience working with individuals with foot and ankle injuries at Mount Sinai.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 80 years old
* Magnetic Resonance Imaging (MRI) confirmed diagnosis of Morton's neuroma - Refractory (greater than 3 month) symptoms to multiple conservative management, including physical therapy, nonsteroidal anti-inflammatory drugs (NSAIDS) and foot orthotics.
* No history of systemic inflammatory conditions such as rheumatoid arthritis
* Able to give written informed consent - Subject has been on a stable dose of analgesic mediation (or not on analgesic medication) for at least 3 weeks and is agreeable to remaining on current regimen for the duration of the study.

Exclusion Criteria:

* Diagnosed complex regional pain syndrome (CRPS)
* Pregnancy - History of intolerance, hypersensitivity or known allergy to lidocaine - Recent history of recent surgical intermetatarsal neuronectomy (within previous 6 months) - Coagulation disorder - Current infection
* Intermetatarsal bursitis
* Metatarsophalangeal joint instability/capsulitis
* Metatarsal stress fracture
* Lumbar radiculopathy
* Tarsal tunnel syndrome
* Frieberg's infraction
* Painful callosities associated with toe deformities
* Peripheral neuropathy
* Diabetes mellitus and peripheral vascular diseases
* Insufficient command of English to complete self-¬report instruments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | up to 12 weeks

SECONDARY OUTCOMES:
Lower extremity functional scale (LEFS) | up to 12 weeks
  A 20-item instrument current level of difficulty with each activity. All 20 items are scored with a maximum score 4 for each item. Scoring ranges from 0-80. The lower the score the higher the disability.

CONTACTS AND LOCATIONS:
Overall Officials: David Spinner, DO, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller, SJ, Nakra, A. Morton's neuroma. In McGlamry's Comprehensive Textbook of Foot and Ankle Surgery, 231-252, Lippincott, Williams, &Wilkins, New York, 2001
- [Background] Peters PG, Adams SB Jr, Schon LC. Interdigital neuralgia. Foot Ankle Clin. 2011 Jun;16(2):305-15. doi: 10.1016/j.fcl.2011.01.010. PMID 21600450
- [Background] Thomson CE, Gibson JN, Martin D. Interventions for the treatment of Morton's neuroma. Cochrane Database Syst Rev. 2004;2004(3):CD003118. doi: 10.1002/14651858.CD003118.pub2. PMID 15266472
- [Background] Okafor B, Shergill G, Angel J. Treatment of Morton's neuroma by neurolysis. Foot Ankle Int. 1997 May;18(5):284-7. doi: 10.1177/107110079701800507. PMID 9167928
- [Background] Coughlin MJ, Pinsonneault T. Operative treatment of interdigital neuroma. A long-term follow-up study. J Bone Joint Surg Am. 2001 Sep;83(9):1321-8. PMID 11568193
- [Background] Lee KT, Kim JB, Young KW, Park YU, Kim JS, Jegal H. Long-term results of neurectomy in the treatment of Morton's neuroma: more than 10 years' follow-up. Foot Ankle Spec. 2011 Dec;4(6):349-53. doi: 10.1177/1938640011428510. Epub 2011 Dec 1. PMID 22134434
- [Background] Su E, Di Carlo E, O'Malley M, Bohne WH, Deland JT, Kennedy JG. The frequency of digital artery resection in Morton interdigital neurectomy. Foot Ankle Int. 2006 Oct;27(10):801-3. doi: 10.1177/107110070602701008. PMID 17054881
- [Background] Tomasian A, Wallace A, Northrup B, Hillen TJ, Jennings JW. Spine Cryoablation: Pain Palliation and Local Tumor Control for Vertebral Metastases. AJNR Am J Neuroradiol. 2016 Jan;37(1):189-95. doi: 10.3174/ajnr.A4521. Epub 2015 Oct 1. PMID 26427837
- [Background] Hegg RM, Kurup AN, Schmit GD, Weisbrod AJ, Atwell TD, Olivier KR, Moynihan TJ, Callstrom MR. Cryoablation of sternal metastases for pain palliation and local tumor control. J Vasc Interv Radiol. 2014 Nov;25(11):1665-70. doi: 10.1016/j.jvir.2014.08.011. Epub 2014 Sep 23. PMID 25255705
- [Background] Prologo JD, Passalacqua M, Patel I, Bohnert N, Corn DJ. Image-guided cryoablation for the treatment of painful musculoskeletal metastatic disease: a single-center experience. Skeletal Radiol. 2014 Nov;43(11):1551-9. doi: 10.1007/s00256-014-1939-x. Epub 2014 Jun 28. PMID 24972918
- [Background] Caporusso EF, Fallat LM, Savoy-Moore R. Cryogenic neuroablation for the treatment of lower extremity neuromas. J Foot Ankle Surg. 2002 Sep-Oct;41(5):286-90. doi: 10.1016/s1067-2516(02)80046-1. PMID 12400711
- [Background] Campos NA, Chiles JH, Plunkett AR. Ultrasound-guided cryoablation of genitofemoral nerve for chronic inguinal pain. Pain Physician. 2009 Nov-Dec;12(6):997-1000. PMID 19935984
- [Background] Connelly NR, Malik A, Madabushi L, Gibson C. Use of ultrasound-guided cryotherapy for the management of chronic pain states. J Clin Anesth. 2013 Dec;25(8):634-6. doi: 10.1016/j.jclinane.2013.05.011. Epub 2013 Aug 27. PMID 23988804
- [Background] Bridges D, Thompson SW, Rice AS. Mechanisms of neuropathic pain. Br J Anaesth. 2001 Jul;87(1):12-26. doi: 10.1093/bja/87.1.12. No abstract available. PMID 11460801
- [Background] Wall PD, Gutnick M. Ongoing activity in peripheral nerves: the physiology and pharmacology of impulses originating from a neuroma. Exp Neurol. 1974 Jun;43(3):580-93. doi: 10.1016/0014-4886(74)90197-6. No abstract available. PMID 4827166
- [Background] Amir R, Michaelis M, Devor M. Membrane potential oscillations in dorsal root ganglion neurons: role in normal electrogenesis and neuropathic pain. J Neurosci. 1999 Oct 1;19(19):8589-96. doi: 10.1523/JNEUROSCI.19-19-08589.1999. PMID 10493758
- [Background] Matzner O, Devor M. Hyperexcitability at sites of nerve injury depends on voltage-sensitive Na+ channels. J Neurophysiol. 1994 Jul;72(1):349-59. doi: 10.1152/jn.1994.72.1.349. PMID 7965019
- [Background] Han KR, Kim C, Chae YJ, Kim DW. Efficacy and safety of high concentration lidocaine for trigeminal nerve block in patients with trigeminal neuralgia. Int J Clin Pract. 2008 Feb;62(2):248-54. doi: 10.1111/j.1742-1241.2007.01568.x. Epub 2007 Nov 23. PMID 18036166